CLINICAL TRIAL: NCT07137858
Title: Adebrelimab Combined With Carboplatin and Albumin-bound Taxanol in the Treatment of Resectable Locally Advanced Oral Squamous Cell Carcinoma Cardiac, Randomized, Phase II Exploratory Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2025-487-02
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC); Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-distance group (Experimental): Each treatment course lasts for three weeks. On the first day of each three-week period, albumin-bound paclitaxel 260mg/m2, carboplatin AUC=5 and adebrelimab 1200mg were administered intravenously. Two treatment courses were carried out in total, and surgery was performed 21 days after the end of the second course of medication. Postoperative radiotherapy and chemotherapy were administered based on the pathological stage. Patients who did not require radiotherapy received adebrelimab (PD-L1 inhibitor) monotherapy maintenance. Patients who required radiotherapy and chemotherapy received monotherapy maintenance during the same period. The duration of medication for all patients was one year (from the first medication time at the initial diagnosis to the last medication time after surgery).
  Interventions: Drug: Preoperative neoadjuvant immunotherapy chemotherapy; Drug: Two courses of preoperative neoadjuvant immunotherapy chemotherapy
- Long-distance group (Active Comparator): Each treatment course lasts for three weeks. On the first day of each three-week period, albumin-bound paclitaxel 260mg/m2, carboplatin AUC=5 and adebrelimab 1200mg are administered intravenously. This treatment is carried out for a total of three cycles, and surgery is performed 21 days after the end of the third cycle. Post-surgery, radiotherapy and chemotherapy are administered based on the pathological stage. Patients who do not require radiotherapy receive adebrelimab (PD-L1 inhibitor) monotherapy maintenance. Patients who require radiotherapy and chemotherapy receive monotherapy maintenance simultaneously. The duration of medication for all patients is one year (from the first administration after diagnosis to the last administration after surgery).
  Interventions: Drug: Preoperative neoadjuvant immunotherapy chemotherapy; Drug: Three courses of preoperative neoadjuvant immunotherapy chemotherapy

INTERVENTIONS:
Drug: Preoperative neoadjuvant immunotherapy chemotherapy — Each treatment course lasts for three weeks. On the first day of each three-week period, albumin-bound paclitaxel 260mg/m2, carboplatin AUC=5 and adalimumab 1200mg are administered intravenously. According to the allocation to the short-course group or long-course group, two or three cycles are carried out respectively, and surgery is performed 21 days after the end of the last cycle of medication. Post-surgery, radiotherapy and chemotherapy are administered based on the pathological stage. Patients who do not require radiotherapy receive maintenance therapy with PD-L1 inhibitor (adalimumab) alone. Patients who require radiotherapy and chemotherapy receive maintenance therapy with the drug alone at the same time. The duration of medication for all patients is one year (calculated from the time of the first medication at the initial diagnosis to the last medication after the surgery).
Drug: Two courses of preoperative neoadjuvant immunotherapy chemotherapy — Each treatment course lasts for three weeks. On the first day of each three-week period, albumin-bound paclitaxel 260mg/m2, carboplatin AUC=5 and adebrelimab 1200mg were administered intravenously. Two treatment courses were carried out in total, and surgery was performed 21 days after the end of the second course of medication. Postoperative radiotherapy and chemotherapy were administered based on the pathological stage. Patients who did not require radiotherapy received adebrelimab (PD-L1 inhibitor) monotherapy maintenance. Patients who required radiotherapy and chemotherapy received monotherapy maintenance during the same period. The duration of medication for all patients was one year (from the first medication time at the initial diagnosis to the last medication time after surgery).
  Arms: Short-distance group
Drug: Three courses of preoperative neoadjuvant immunotherapy chemotherapy — Each treatment course lasts for three weeks. On the first day of each three-week period, albumin-bound paclitaxel 260mg/m2, carboplatin AUC=5 and adebrelimab 1200mg are administered intravenously. This treatment is carried out for a total of three cycles, and surgery is performed 21 days after the end of the third cycle. Post-surgery, radiotherapy and chemotherapy are administered based on the pathological stage. Patients who do not require radiotherapy receive adebrelimab (PD-L1 inhibitor) monotherapy maintenance. Patients who require radiotherapy and chemotherapy receive monotherapy maintenance simultaneously. The duration of medication for all patients is one year (from the first administration after diagnosis to the last administration after surgery).
  Arms: Long-distance group

SUMMARY:
Neoadjuvant immunochemotherapy can effectively increase the postoperative pathological complete response rate, improve the survival rate of patients, and reduce the risk of recurrence in oral squamous cell carcinoma (OSCC). Programmed death ligand-1 (PD-L1) plays a role in inhibiting the cancer-immune cycle by binding to negative regulatory factors of T cell activation such as PD-1 and B7.1. It has achieved good therapeutic effects in lung cancer, liver cancer and other cancers. Previous studies have shown that three cycles of PD-L1 inhibitors combined with chemotherapy have satisfactory efficacy and safety in locally advanced oral squamous cell carcinoma. However, during the three-cycle treatment process, due to the accumulation of drug toxicity, patients' tolerance to adverse reactions decreases, increasing the risk of serious adverse events and psychological pressure on patients. Based on this, this study aims to explore the efficacy of two cycles of avelumab (PD-L1 inhibitor) combined with chemotherapy in locally advanced oral squamous cell carcinoma, to explore whether it can achieve the same efficacy as three cycles while shortening the treatment time, reduce the risk of serious adverse events, and further verify the efficacy and safety of PD-L1 inhibitors combined with chemotherapy in the treatment of locally advanced oral squamous cell carcinoma. This study uses the postoperative pathological complete response (PCR) rate as the primary outcome indicator, and the objective response rate (ORR), major pathological response (MPR) rate, 2-year disease-free survival (EFS) rate, and 2-year and 5-year overall survival (OS) rate as secondary outcome indicators to evaluate the efficacy and long-term survival impact.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old;
2. According to the 8th edition guidelines of the American Joint Committee on Cancer (AJCC), patients with pathologically confirmed head and neck squamous cell carcinoma (oral cavity including cheek, tongue, gum, floor of mouth, palate, maxillary sinus), and having stage III-IVB tumors other than oropharyngeal cancer;
3. Before enrollment, the resectable tumors were evaluated by head and neck surgeons, and clinical evidence of distant metastasis was excluded;
4. According to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, at least one measurable tumor lesion was present;
5. The performance status of the Eastern Cooperative Oncology Group (ECOG) was 0-1;
6. Blood routine: White blood cell count (WBC) ≥ 3.0×109/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet (PLT) ≥ 100×109/L; Hemoglobin level (HGB) ≥ 9.0 g/dL (without corresponding supportive treatments such as blood transfusion and increase in white blood cells within 7 days);
7. Liver function: For patients without liver metastasis, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); Albumin (ALB) ≥ 30 g/L;
8. Renal function: Serum creatinine ≤ 1.5 times ULN or creatinine clearance rate (CrCl) ≥ 50 mL/min (using the Cockcroft/Gault formula); Urinary protein (UPRO) < (++), or 24-hour urine protein quantity < 1.0 gram;
9. HPV status of oropharyngeal cancer was determined by p16 IHC. If more than 70% of tumor cells showed strong diffuse nuclear and cytoplasmic staining, the sample was considered p16 positive;
10. Within the past 30 days, no other clinical trial projects were participated in;
11. Patients who voluntarily participated in this project and signed the informed consent form.

Exclusion Criteria:

1. The patient's blood indicators were abnormal, and their liver and kidney functions were also abnormal. After a multidisciplinary consultation, it was determined that they could not tolerate the process of this clinical study.
2. The patient had previously suffered from tumors in other parts of the body, or had undergone anti-tumor treatments such as surgery, chemotherapy, and radiotherapy in the past.
3. Due to personal, social, or economic reasons, they were unable to complete the entire clinical study process.
4. The patient had previously suffered from severe systemic diseases that could not be cured or controlled by medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pathological complete response rate | All patients were treated within 7 working days after surgery
  There were no residual tumor cells in the pathological sections of the surgically resected primary lesion and lymph node specimens. The main judgment method is that the postoperative specimen is sent to the pathology department for fixation, sectioning, and observation. Two pathologists read the images to determine whether the tumor was residual. If there was any disagreement between them, the third senior pathologist would discuss and decide.

SECONDARY OUTCOMES:
Major pathological response rate | All patients were treated within 7 working days after surgery
  Proportion of patients with 10% or less viable tumor cells in the primary lesion specimen.
Objective tumor response rate | All patients were treated 21 days after the last dose of preoperative neoadjuvant immunochemotherapy
Event-free survival at 2 years | Within 2 years after completion of all treatments
The overall survival rates for 2 years and 5 years | Within the next 2 years and 5 years after all treatments are completed

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT07137858/Prot_SAP_ICF_000.pdf